CLINICAL TRIAL: NCT03554655
Title: The Momentum Trial: The Efficacy of Using a Smartphone Application to Support Shared Decision Making Through Patient Activation in People With a Diagnosis of Schizophrenia in Outpatient Treatment Settings
Brief Title: The Efficacy of Using a Smartphone App to Support Shared Decision Making in People With a Diagnosis of Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: TrygFonden, Denmark (Industry); Odense Patient Data Explorative Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 115441; H-17025550 (Other: Regional Ethics Committee in The Capital Region of Denmark)
Record Dates: First submitted 2018-04-30; First posted 2018-06-13 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia, Schizotypal and Delusional Disorders
Keywords: Shared decision making; Patient activation; Schizophrenia; First-episode psychosis; mHealth; Randomized clinical trial
MeSH Terms: conditions — Schizophrenia; Schizophrenia, Paranoid; Patient Participation

STUDY DESIGN:
Intervention Model Description: A two-arm, observer-blinded, parallel group randomised controlled superiority trial will be used for this intervention. Participants will be placed in one of two groups: Intervention group: treatment as usual (TAU) together with the Momentum app or (2) Control group: TAU without the Momentum app.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Given the nature of the intervention, patients and healthcare providers cannot be kept blinded. Investigators responsible for data collection and data entry will be blinded as to patient allocation until all outcomes have been collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Momentum app (Experimental): Intervention Group will receive treatment as usual together with the Momentum app.
  Interventions: Device: Momentum app
- Control (No Intervention): Control Group will receive treatment as usual without the Momentum app.

INTERVENTIONS:
Device: Momentum app — The Momentum system consists of a smartphone app (for the patient) and a web portal (for the provider). Information entered in the app by the patient will automatically be transferred to the web portal for the provider to see. While one goal of the system is to support SDM, the Momentum app is not a classic decision aid focusing on finding a choice to a one-off treatment decision. Instead, the Momentum app is an aid to support some of the underlying elements behind SDM such as collaboration with one's provider, awareness and eliciting of one's needs, preferences and values.
  Arms: Intervention: Momentum app

SUMMARY:
This study investigates the effects of using a smartphone app to support shared decision making (SDM) for people with schizophrenia-spectrum disorders in an outpatient treatment setting. Patients are randomized to specialized early intervention treatment with the Momentum app or without the app. The primary objective is to investigate the effect of the app on patient activation 6 months after baseline. Secondary outcomes are positive and negative symptoms, level of functioning; working alliance; self-efficacy; treatment satisfaction; hope; level of SDM; and perceived efficacy in patient-provider interaction. Explorative outcomes are self-perceived usefulness of the Momentum app.

DETAILED DESCRIPTION:
Background:

Shared decision making (SDM) may be associated with positive health outcomes for the patient. While practitioners provide a professional expertise with information on the diagnosis, course of the illness, treatment options and potential side effects, patients are experts on their own needs, treatment preferences and goals. In mental healthcare, SDM have been assessed as a promising treatment intervention to promote patient involvement and clinical guidelines advocate the use of SDM as a patient-centered mental health care and a mean to increase patient empowerment. Although SDM today seems to be a preferred model for clinical decision-making for both patients and providers in mental health, patients indicate that they are not involved as much as they want to be in their treatment. Studies on SDM interventions for people with mental health issues are somewhat sparse and due to a small number of RCT studies, the evidence on SDM in mental health has been concluded as encouraging but inconclusive.

Based on recent research, a digital healthcare solution which links patients and providers together could assist in providing support and potentially promote SDM. Findings from existing randomized controlled trials suggest that electronic aids to support SDM are a promising mean to engage patients in their mental health treatment. Recent systematic reviews do, however, highlight a need for more evidence-based research on the efficacy and effectiveness of mental health apps.

Intervention:

Momentum is a smartphone app, developed to support people with schizophrenia-spectrum disorders to prepare for treatment consultations while becoming more involved in treatment decisions. The app was developed in the period of 2013-2014 to support SDM in the Mental Health Services of the Capital Region of Denmark in a process of co-creation. Afterwards, the app was tested by 116 mental health professionals and 78 patients from three different mental health treatment sites: community of mental health, inpatient- and outpatient treatment sites. The app has since then been optimized based on the feedback received from the study participants.

Aim:

The purpose of this trial is to investigate the effects of the smartphone app Momentum for people with a diagnosis of schizophrenia, schizotypal or delusional disorders within outpatient treatment settings in a randomized design. Our main hypothesis is that patients using the Momentum app in combination with receiving specialized early intervention treatment (i.e. treatment as usual (TAU)), compared to patients only receiving TAU, will show greater improvements in patient activation, 6 months after baseline (primary outcome). Our secondary hypothesis is that patients using the Momentum app in combination with receiving TAU, compared to patients only receiving TAU, will show greater improvements regarding self-perceived level of SDM; self-efficacy; the therapeutic alliance; hope and optimism; satisfaction with treatment; patient's confidence in communicating preferences and concerns to their provider; severity of symptoms and; level of functioning (secondary outcomes). Lastly, the investigators hypothesize that there is a correlation between the effects of using the Momentum app and self-reported usefulness of the Momentum app and/or app usage (user sessions per day, screen views per day, screens per session, session duration and session instances, user retention) (explorative outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Adults of both sexes aged 18+
* A diagnosis of schizophrenia, schizotypal or delusional disorder (ICD-10 codes: F20-F29)
* The patient have received treatment for a maximum of 18 months at the start of the intervention from one of five participating OPUS centre in the Mental Health Services of the Capital Region of Denmark

Exclusion Criteria:

* Do not understand or speak Danish
* Unable to give written informed consent to participate in the trial at the described terms
* Are participating in other research studies involving OPUS treatment and an app
* Do not have daily access to a smartphone
* Are suffering of mental retardation or dementia (F. 70-F.79, F.00-F.03)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 194 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Change in patient activation measured with the Consumer Health Activation Index - Mental Health (CHAI-MH) | baseline, 3 months and end of intervention (6 months)
  Completed by patients. The 10-item instrument was developed based on 5 key domains: knowledge, self-efficacy, motivation and beliefs, actions, and internal locus of control. The questionnaire is rated on a 6-point Likert scale ranging from "Strongly disagree" to "Strongly agree". Afterwards, the scores are transformed into a theoretical value from 0 to 100, with higher scores signifying a stronger involvement in the treatment and confidence in the ability to take care of one's own health and health treatment.

SECONDARY OUTCOMES:
Change in self-efficacy measured with the General Self-Efficacy scale (GSE) | baseline, 3 months and end of intervention (6 months)
  Completed by patients. The questions consists of 10 items rated on a 4-point Likert scale ranging from "not at all true" (1) to "exactly true" (4) with higher scores indicating higher self-efficacy.
Change in preparedness for decision making measured with the scale Preparation for Decision Making (PrepDM) | baseline and 6 months
  Completed by patients. The 10-item instrument measures the patient's perception of how useful a decision aid or other decision support intervention is. The questionnaire is rated on a 5-point Likert scale from "Not at all" (1) to "A great deal" (5) with higher scores indicating a higher level of preparedness to communicate with one's care provider regarding health decisions.
Change in hope measured with the Adult State Hope Scale (ASH) | baseline, 3 months and end of intervention (6 months)
  Completed by patients. The 6-item instrument is rated on a Likert-scale from 1-8, with higher scores indicating higher levels of hope.
Change in the efficacy of interactions measured with the scale Perceived Efficacy in Patient-Provider Interactions (PEPPI) | baseline, 3 months and end of intervention (6 months)
  Completed by patients. The 5-item instrument measures the assessment of patient's confidence in communicating with their physician. The questionnaire is rated on a 10-point Likert scale, with higher scores indicating higher perceived efficacy in the interactions
Change in treatment satisfaction measured with the Client Satisfaction Questionnaire (CSQ) | baseline and 6 months
  Completed by patients. The 8-item instrument measures a patient's satisfaction with treatment. Each item is scored on a 4-point Likert scale, with higher scores indicating higher satisfaction.
App Rating Questionnaire (ARQ) and usage of the Momentum app will be combined to report patients self-perceived usefulness of the app | 6 months
  Completed by patients in the intervention Group. ARQ is used to measure the users experience with the app. Higher scores indicating higher perceived usefulness of the app.
Change in treatment alliance measured with the Working Alliance Inventory - short version (WAI-S). Patient version. | baseline and 6 months
  Completed by patients. The questionnaire consists of 12 items rated on a 7-point Likert scale, with higher scores indicating better self-perceived working alliance with ones provider.
Change in treatment alliance measured with the Working Alliance Inventory - short version (WAI-S). Clinician version. | baseline and 6 months
  Completed by providers.The questionnaire consists of 12 items rated on a 7-point Likert scale, with higher scores indicating better self-perceived working alliance with ones patient.
Clinical Decision Making Style - Service user (CDMS-P) | baseline
  Completed by patients. The 21-item measures preferences in clinical decision making. The questionnaire is rated on a 5-point Likert scale with higher scores indicating a higher desire to be an active participant in decision making and to be provided with information.
Clinical Decision Making Style - Staff questionnaire (CDMS-S). | baseline
  Completed by providers. The questionnaire is rated on a 5-point Likert scale with higher scores indicating a higher desire by the clinician for active service user participation in decision making and to provide information to the service user.
Service Engagement Scale - Collaboration sub-domain only (SES) | baseline and 6 months
  Completed by providers. The scale is a 14-item measurement for the provider to rate their patient's engagement level on the subscale Collaboration. Each item is scored on a 4 point Likert scale, with higher scores indicating poorer engagement.
Change in positive symptoms measured by the Scale for the Assessment of Positive Symptoms (SAPS) | baseline and 6 months
  Each dimension within SAPS is scored between 0-5 with higher scores indicating higher symptom severity
Change in negative symptoms measured by the Scale for the Assessment of Negative Symptoms (SANS) | baseline and 6 months
  Each dimension within SANS is scored between 0-5 with higher scores indicating higher symptom severity
Change in level of functioning measured with the Global Assessment of Functioning (GAF) | baseline and 6 months
  GAF assesses a person's psychosocial functioning (scores 1-100), with higher scores indicating a higher functioning level.
Change in level of functioning measured with the Personal and Social Performance Scale (PSP) | baseline and 6 months
  PSP assesses a person's functioning level within four domains; socially useful activities; Personal and social relationships; Self-care; Disturbing and aggressive behaviors. PSP is scored 1-100, with higher scores indicating a higher functioning level.

OTHER OUTCOMES:
Objective data on app usage | 3 months and 6 months
  Objective data covers: user sessions per day, screen views per day, screens per session, session duration and session instances, user retention
Anti-psychotic medicine | baseline and 6 months
  Use and adherence of anti-psychotic medicine
Adherence to treatment | baseline, 3 months and 6 months
  number of no-shows to treatment consultations compared to number of planned consultations
Hospital admissions | baseline, 3 months and 6 months
  Number of hospital admissions

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Korsbek, ph.d., Principal Investigator — Mental Health Services in the Region of Southern Denmark, Odense
Locations (7):
- Denmark (7):
  - OPUS Amager, Amager
  - OPUS Ballerup, Ballerup Municipality
  - OPUS Glostrup, Brøndby
  - OPUS Hvidovre, Brøndby
  - OPUS Valby, Brøndby
  - OPUS Hillerød, Hillerød
  - OPUS Østerbro, København Ø

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vitger T, Hjorthoj C, Austin SF, Petersen L, Tonder ES, Nordentoft M, Korsbek L. A Smartphone App to Promote Patient Activation and Support Shared Decision-making in People With a Diagnosis of Schizophrenia in Outpatient Treatment Settings (Momentum Trial): Randomized Controlled Assessor-Blinded Trial. J Med Internet Res. 2022 Oct 26;24(10):e40292. doi: 10.2196/40292. PMID 36287604
- [Derived] Vitger T, Austin SF, Petersen L, Tonder ES, Nordentoft M, Korsbek L. The Momentum trial: the efficacy of using a smartphone application to promote patient activation and support shared decision making in people with a diagnosis of schizophrenia in outpatient treatment settings: a randomized controlled single-blind trial. BMC Psychiatry. 2019 Jun 17;19(1):185. doi: 10.1186/s12888-019-2143-2. PMID 31208376
- See also: OPEN — https://open.rsyd.dk/OpenProjects/openProject.jsp?lang=da&openNo=451